CLINICAL TRIAL: NCT04394832
Title: Reducing Intrusive Memories of Trauma Using a Visuospatial Interference Intervention With Refugees With Posttraumatic Stress Disorder (PTSD): A Pilot Study
Brief Title: Reducing Intrusive Memories in Refugees and Asylum Seekers With PTSD: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: University of Surrey (Other)
Collaborators: Central and North West London NHS Foundation Trust (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPON 2019 032 FHMS (A)
Record Dates: First submitted 2020-04-21; First posted 2020-05-19 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Mental Disorder; Trauma and Stressor Related Disorders
Keywords: Intrusive Memories; Post-Traumatic Stress Disorder; Cognitive Task Interference
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Mental Disorders; Trauma and Stressor Related Disorders

STUDY DESIGN:
Intervention Model Description: Multiple baseline case-series design (AB), with a randomised duration of baseline length.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baseline phase, followed by intervention phase (Experimental): Within the baseline phase, measurements of the primary outcome measure (frequency of intrusive memories of trauma) were collected in a pen-and-paper diary for up to three weeks (dependent on baseline length). Individual baseline phases will be used as control periods.
  In the intervention phase the participant was offered around five intervention sessions with a researcher. Each session the participant chose which intrusive memory they would like to focus on and the cognitive task was completed. The intervention included a memory reminder cue, a 10-minute time gap and then around 20 minutes playing the mobile phone game Tetris, using mental rotation instructions. Participants were given instructions to continue to use the technique self-guided in the subsequent week. Measurements of the primary outcome measure (frequency of intrusive memories of trauma) were collected in a pen-and-paper diary.
  Interventions: Behavioral: Brief cognitive intervention

INTERVENTIONS:
Behavioral: Brief cognitive intervention — See the information provided in the experimental arm description.

SUMMARY:
This research study was designed to investigate the use of a simple cognitive task for decreasing the number of intrusive memories of traumatic events experienced by refugees and asylum seekers with a diagnosis of Post-traumatic Stress Disorder (PTSD) currently living in the UK. The intervention included a memory reminder cue, a 10-minute time gap and then around 20 minutes playing the mobile phone game Tetris, using mental rotation instructions. The study had a multiple baseline case-series design (AB), with a randomised duration of baseline length up to three weeks. Thus, participants completed a no-intervention phase of up to three weeks, followed by an intervention phase. Please see the intervention section for more details about the intervention sessions. Follow ups were conducted after each week to monitor the frequency of intrusive memories of trauma in a pen-and-paper diary. It was predicted that participants would report fewer intrusive memories after receiving the intervention than in the preceding baseline phase.

DETAILED DESCRIPTION:
The study was conducted at a specialist National Health Service (NHS) mental health service for refugees, asylum seekers and forced migrants suffering from Post-Traumatic Stress Disorder (PTSD). Four participants were enrolled in the study. This was initially intended to be a larger study (n=15) but recruitment stopped due to the COVID-19 pandemic and advice from the trust R&D and NHS service manager that face-to-face appointments should no longer go ahead at the NHS clinical recruitment site. The trust R&D advised that only participants who had started the intervention should continue and only if done remotely. An amendment was approved for remote delivery of the intervention. Two of the four participants who gave informed consent continued to participate in the study. They met with a researcher remotely via video technology. The other two participants instead continued to receive standard care by the NHS service but did not continue with the research study. This study was a pilot.

The study had a multiple baseline case-series design (AB), with a randomised duration of baseline length up to three weeks. At the start of the baseline phase, participants created, with the help of the researcher, a list of their most frequent and distressing intrusive memories of trauma. Each intrusive memory was given a label (for example; a letter, colour or symbol) so that the frequency of each intrusive memory could be monitored in a pen and paper diary. The frequency of specific intrusive memories the person experienced after they had received the intervention will be compared to the frequency of specific intrusive memories they had during the baseline phase. For each specific intrusion, the period prior to that intrusion being targeted in an intervention session was the baseline phase (A); therefore, the baseline phase included the minimum baseline duration (lasting up to three weeks) plus the additional weeks in which the specific intrusion remained untargeted by the intervention. The post intervention phase (B) was the time after the specific intrusion was targeted. Some intrusive memories on the list were not targeted by the intervention but were monitored (through the intrusion diary) throughout the duration of the study for comparison.

This study was a follow-up to a study conducted in Sweden with refugees. ClinicalTrials.gov Identifier: NCT03760601. The research is extending the previous research to refugees and asylum seekers with a diagnosis of PTSD, accessing a secondary care mental health service and living in the United Kingdom (UK).

ELIGIBILITY:
Inclusion Criteria:

* are on the wait list for treatment (trauma focused therapy) at Woodfield Trauma Service
* aged 18-65
* have experienced intrusive memories in the past two weeks, as assessed by scoring 1 or above on question 1 of the PCL-5
* are able to communicate with the researcher, with or without an interpreter
* have a fixed abode. This is operationalised as having a current address (including B&B or open access hostel) and evidence indicating that the person is likely to have a reliable address throughout the study. This is necessary to avoid sample attrition.
* can commit to attending regular appointments and keeping an intrusion diary throughout the duration of the study.

Exclusion Criteria:

* a current diagnosis of schizophrenia or bipolar disorder type 1
* Intelligence Quotient (IQ) < 80
* acute suicide risk
* substance dependence
* have been unable to complete the routine questionnaires given to new patients in the service at assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Frequency of intrusive memories | Daily through study completion, an average of 3 months. Change is assessed from baseline to post-intervention.
  Number of intrusive memories of traumatic events recorded by participants in a pen and and paper diary.

SECONDARY OUTCOMES:
Concentration | Baseline and 2-weeks post-intervention
  A brief bespoke measure of concentration adapted from that used previously with refugees (Holmes et al., 2017). It has three questions about disruption to concentration from intrusive memories. A higher score on each question means a worse outcome.
Social and Occupational Activity Tally (SOAT) | Baseline and 2-weeks post-intervention
  Developed by Woodfield Trauma Service. The measure asks how many hours the person has spent doing various activities in the past two weeks (for example, domestic chores, exercise, cultural activities). A higher score means a better outcome.
Dissociation | Baseline and 2-weeks post-intervention
  Four items from the Dissociative Experiences Scale II - items two, three, 14 and 20 (DES II; Carlson, & Putnam, 1993). Each item asks how often (from 0% to 100% of the time) the dissociative experience described happens to the individual. A higher score on each question means a worse outcome.
Post-Traumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (PCL-5) | Baseline and 2-weeks post-intervention
  The PCL-5 (Weathers, Litz, Keane, Palmieri, Marx, & Schnurr, 2013) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Total scores can range from 0 to 80, with higher scores meaning a worse outcome.
Patient Health Questionnaire (PHQ-9) | Baseline and 2-weeks post-intervention
  The PHQ-9 (Kroenke, Spitzer & Williams, 2001) is a nine-item self-report measure that assesses the nine DSM-IV symptoms of depression. Total scores can range from 0 to 27, with higher scores meaning a worse outcome.
World Health Organisation Disability Assessment Schedule 2.0 (WHO DAS 2.0) 12 item version | Baseline and 2-weeks post-intervention
  The WHO DAS 2.0 (World Health Organisation, 2010) is a measure of health and disability. Total scores can range from 0 to 48, with higher scores meaning a worse outcome.

OTHER OUTCOMES:
Self-Guided Intervention Adherence Questionnaire | Intervention weeks 2-5, 1 week post-intervention and 2 weeks post-intervention
  A bespoke measure to assess adherence to self-guided practice of the intervention. It includes four questions to assess how often, and for how long, the person played Tetris after experiencing intrusive memories during the previous week.
Feedback Questionnaire | 1-week post-intervention.
  A bespoke questionnaire to gain feedback on the intervention. It includes 16 questions to assess acceptability and usefulness of the intervention with a variety of response options including yes/no, visual analogue scales and open responses.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Greenfield, Principal Investigator — University of Surrey
Locations (1):
- Woodfield Trauma Service, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No